CLINICAL TRIAL: NCT07215871
Title: Rechallenge With a Low Pathogenicity Avian H10N7 Influenza Virus in Healthy Human Volunteers Previously Challenged With H10N7 Influenza
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 10002421; 002421-I
Record Dates: First submitted 2025-10-10; First posted 2025-10-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-10-21

CONDITIONS: Influenza Infection; Infections; Respiratory Virus Infections; Respiratory Tract Infections; RNA Viruses; Orthomyxoviridae Infections; Viral Diseases
Keywords: Influenza A; H10N7; Challenge Model; Influenza; Human Challenge
MeSH Terms: conditions — Infections; Respiratory Tract Infections; Orthomyxoviridae Infections; Virus Diseases; Influenza, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- H10N7 Infection (Experimental): Subjects will be infected with H10N7 virus.
  Interventions: Biological: A/Mallard/Ohio-99/MM4/1989 H10N7

INTERVENTIONS:
Biological: A/Mallard/Ohio-99/MM4/1989 H10N7 — Low pathogenicity avian influenza virus H10N7

SUMMARY:
Background:

Influenza (flu) is a virus that can infect humans and animals. In humans, the flu can cause mild symptoms such as fever, cough, sore throat, runny nose, muscle aches, headaches, and fatigue. It can also cause sinus infections or pneumonia. Some flu strains, such as H5N1 and H7N9, which come from birds, can lead to more severe symptoms or death. Others, like H10N7, also come from birds but usually cause mild symptoms. Researchers want to study bird flu in humans to help develop new flu vaccines and treatments.

Objective:

To learn more about how bird flu viruses infect humans.

Eligibility:

Healthy people aged 18 to 55 years who were infected with the H10N7 bird flu strain as part of a previous study.

Design:

Participants who were infected with H10N7 in a previous study will be infected again with the same virus. The virus will be sprayed into their nostrils.

Participants will stay in the hospital for at least 9 days. They will stay in an isolation unit. No outside visitors will be allowed.

During their stay, participants will provide blood, urine, and nasal fluid samples. They will have tests of their heart and lung function. They will complete questionnaires about their symptoms.

Participants will remain in the hospital until they test negative for the flu 2 days in a row. They will continue to complete questionnaires about their symptoms for 2 weeks after they were infected with the virus.

Participants will have 2 follow-up visits, at 5 weeks and 9 weeks after they were infected. They will have a physical exam and provide samples of blood and nasal fluids. They will have a test of their heart function.

DETAILED DESCRIPTION:
This is a single-center study to evaluate infection after a second exposure to a low pathogenicity avian influenza A H10N7. Participants who have previously been challenged with H10N7 willbe rechallenged with 10^7 Tissue Culture Infective Dose (TCID50) virus and followed for a minimum of 9 weeks after inoculation. The study hypothesis is that mild to moderate influenza disease (MMID) can be induced with the A/Mallard/Ohio/99/1989 H10N7 influenza challenge virus on re-exposure despite the potential development of immunity after the last challenge. This will be evaluated by monitoring participants for influenza disease symptoms, viral shedding, and immunological response. The primary way MMID will be determined will be through clinical testing for influenza and symptom monitoring.

Objectives:

Primary Objective:

1. Determine if participants develop MMID after a second challenge with A/Mallard/Ohio/99/1989 H10N7.

Secondary Objectives:

1. Evaluate clinical disease, identify clinical markers, and observe initiation of shedding, length of shedding, and pathogenesis in participants with low pathogenicity avian influenza A infection.
2. Evaluate immune response after a second challenge with H10N7 compared to the initial challenge.

Exploratory Objectives:

1. Evaluate additional host immune responses, viral replication, viral fitness, and intrahost evolution.
2. Evaluate clinical and virologic outcomes as outlined in primary and secondary objectives in subgroups of interest.
3. Determine correlates of protection against H10N7 challenge.

Endpoints:

Primary Endpoint:

1. Rate of MMID, defined as a positive US Food and Drug Administration (FDA)-approved clinical test for influenza plus one or more influenza symptoms.

   Secondary Endpoints:
2. Clinical outcomes after challenge including: a. Mean duration and quantity of shedding of influenza in nasal wash/synthetic absorptive matrices (SAM) by quantitative real-time polymerase chain reaction (PCR).

   b. Mean duration and number of symptoms and signs elicited by daily oral history and clinical exam compared to prior infection.

   c. Mean daily and total score of influenza patientreported outcome (FLU-PRO) questionnaire.
3. Immunological responses after challenge including:

   1. Serum hemagglutination (HA) inhibition (HAI) and/or enzyme-linked immunosorbent assay (ELISA) against HA.
   2. Serum neuraminidase (NA) inhibition (NAI) and/or ELISA titers against NA.
   3. Mucosal ELISA titers against HA and NA.

Exploratory Endpoints:

1. Immune response and viral factors including:

   1. Levels and type of influenza infection induced gene expression determined by human gene expression analysis and high-throughput sequencing.
   2. Characterization of B- and T-cell responses.
   3. Change in viral genotype from the inoculum of virus isolated from infected participants.
2. MMID, shedding, symptom rates, and immune responses in subgroups of interest (including but not limited to those who

   had/had not MMID after the first challenge, had/had not shedding after first challenge).
3. Immunological correlates of protection (like HAI, NAI, mucosal responses, cellular responses) in protecting against clinical outcomes (including MMID, shedding, symptoms).

ELIGIBILITY:
* INCLUSION CRITERIA:

An individual must meet all of the following criteria to be eligible for study participation:

1. Previously participated in the H10N7 influenza challenge study 20-I-0160 ("Dose- Escalation Study of a Low Pathogenicity Avian H10N7 Influenza Virus in a Healthy Human Challenge Model") and given a viral challenge H10N7.
2. >=18 and <=55 years of age.
3. Able to provide informed consent.
4. Agrees to not use tobacco products, marijuana, or vaping products through the last mandatory visit.
5. Willing to remain in isolation for a minimum of 9 calendar days (or for the duration of viral shedding) and to comply with all study requirements.
6. A male subject is eligible for the study if he meets one of the following criteria, beginning at least 4 weeks prior to enrollment and continuing until follow-up visit #2:

   1. Is infertile, including history of successful vasectomy.
   2. Agrees to practice abstinence.
   3. Agrees that, with heterosexual intercourse with a fertile female partner, he will use a condom with spermicide and his female partner will use an acceptable form of contraception (see inclusion criterion 7c).
7. A female participant is eligible for this study if she is not pregnant or breastfeeding and meets one of the following criteria, beginning at least 4 weeks prior to enrollment and continuing until follow-up visit #2:

   1. Is infertile, including postmenopausal status (as defined by no menses for >=1 year) or history of hysterectomy.
   2. Agrees to practice abstinence.
   3. Agrees that, with heterosexual intercourse with a fertile male partner, she will use an acceptable form of contraception, and her male partner will use a condom with spermicide. Acceptable effective methods of female contraception include the following: bilateral tubal ligation, implant of levonorgestrel, injectable progestogen, intrauterine device, oral contraceptive pills, and diaphragm with spermicide.
8. Willing to have samples stored for future research.
9. Human immunodeficiency virus (HIV) uninfected with a negative test within 90 days of inoculation (Day 0).
10. Ability to speak English.

EXCLUSION CRITERIA:

An individual meeting any of the following criteria will be excluded from study participation:

1. Has self-reported or medically documented significant medical condition including but not limited to:

   1. Chronic pulmonary disease (e.g., asthma, emphysema).
   2. Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
   3. Chronic medical conditions requiring close medical follow-up or hospitalization during the past 5 years (e.g., insulin-dependent diabetes mellitus, renal dysfunction, hemoglobinopathies).
   4. Immunosuppression or ongoing malignancy.
   5. Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
   6. Post-infectious or post-vaccine neurological sequelae.
2. Has close or household (i.e., share the same apartment or house) high-risk contacts including but not limited to:

   1. Persons >=65 years of age.
   2. Children <=5 years of age.
   3. Residents of nursing homes.
   4. Persons of any age with significant chronic medical conditions such as:

      * Chronic pulmonary disease (e.g., asthma).
      * Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
      * Chronic medical conditions requiring medical follow-up or hospitalization during the past 5 years (e.g., insulin-dependent diabetes mellitus, renal dysfunction, hemoglobinopathies).
      * Immunosuppression or cancer.
      * Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
      * Persons who are receiving long-term aspirin therapy.
      * Women who are pregnant, trying to become pregnant, or breastfeeding.
3. Has a body mass index (BMI) <=18.5 or >=35.
4. Smokes more than 4 cigarettes or other tobacco products on a weekly basis or any type of vaping/e-cigarette use more than 4 times per week.
5. History of facial reconstructive procedures or nasopharyngeal malformation that would preclude nasal sampling.
6. Positive for hepatitis B or hepatitis C infections.
7. Complete blood count (CBC) with differential outside of the NIH Department of Laboratory Medicine (DLM) normal reference range and deemed clinically significant by the PI.
8. Grade 2 or higher hemoglobin decrease for female participants or Grade 1 or higher hemoglobin decrease for male participants.
9. Chemistries in the acute care, mineral, and/or hepatic panels, and/or any of the following: lactate dehydrogenase (LDH), uric acid, creatine kinase, and total protein outside of the NIH DLM normal reference range and deemed clinically significant by the PI.
10. Urinalysis outside of the NIH DLM normal reference range and deemed clinically significant by the PI.
11. Clinically significant abnormality as deemed by the PI on ECG.
12. Clinically significant abnormality as deemed by the PI on ECHO.
13. Clinically significant abnormality as deemed by the PI on the PFT and/or spirometry.
14. Recent acute illness within 1 week of admission to the NIH CC.
15. Positive test for any respiratory virus on nasal wash (including but not limited to SARSCoV-2) on admission.
16. Known allergy to any component of the interventional agent.
17. Known allergy to treatments for influenza (including but not limited to oseltamivir, nonsteroidals anti-inflammatory drugs).
18. Known allergy to 2 or more classes of antibiotics (e.g., penicillins, cephalosporins, fluoroquinolones, or glycopeptides).
19. Receipt of influenza vaccine within 8 weeks prior to enrollment.
20. Receipt of a broadly protective influenza vaccine or avian influenza vaccine.
21. Natural infection with avian influenza outside of the research setting.
22. Having influenza infection within 8 weeks prior to enrollment.
23. Receipt of blood or blood products (including immunoglobulins) within 3 months prior to enrollment.
24. Receipt of any unlicensed drug within 3 months or 5.5 half-lives (whichever is greater) prior to enrollment.
25. Receipt of any unlicensed vaccine within 6 months prior to enrollment.
26. Self-reported or known history of current alcoholism or drug abuse, or positive urine/serum test for drugs of abuse (i.e., amphetamines, cocaine, benzodiazepines, opiates, or metabolite and tetrahydrocannabinol or metabolites).
27. Self-reported or known history of psychiatric or psychological issues deemed by the PI to be a contraindication to protocol participation.
28. Known close contact with anyone known to have influenza in the past 7 days.
29. Known close contact with anyone known to have COVID-19 in the past 14 days.
30. History of COVID-19-related complications, including, but not limited to: inpatient hospitalization, required the use of oxygen, and/or on-going sequelae.
31. Any condition that, in the judgment of the PI, is a contraindication to protocol participation or impairs the volunteer s ability to give informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-09-29 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Determine if participants develop mild-to-moderate influenza disease after a second challenge with H10N7. | 9 days
  Subjects will remain inpatient for 9 days total to evaluate for infection and symptoms after infection with H10N7.

SECONDARY OUTCOMES:
Evaluate clinical disease, identify clinical markers, and observe initiation of shedding, length of shedding, and pathogenesis in participants with low pathogenicity avian influenza A infection. | 3 months
  Subjects will be evaluated for clinical disease, shedding and analysis will be done on these findings compared to shedding after infection with H10N7 a second time.
Evaluate immune response after a second challenge with H10N7 compared to the initial challenge. | 2 years
  We will conduct laboratory evaluation of antibody levels to the H10N7 virus compared to first challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Luca T Giurgea, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi YS, Baek YH, Kang W, Nam SJ, Lee J, You S, Chang DY, Youn JC, Choi YK, Shin EC. Reduced antibody responses to the pandemic (H1N1) 2009 vaccine after recent seasonal influenza vaccination. Clin Vaccine Immunol. 2011 Sep;18(9):1519-23. doi: 10.1128/CVI.05053-11. Epub 2011 Aug 3. PMID 21813667
- [Background] Memoli MJ, Han A, Walters KA, Czajkowski L, Reed S, Athota R, Angela Rosas L, Cervantes-Medina A, Park JK, Morens DM, Kash JC, Taubenberger JK. Influenza A Reinfection in Sequential Human Challenge: Implications for Protective Immunity and "Universal" Vaccine Development. Clin Infect Dis. 2020 Feb 14;70(5):748-753. doi: 10.1093/cid/ciz281. PMID 30953061
- [Background] Skowronski DM, Li Y, Tweed SA, Tam TW, Petric M, David ST, Marra F, Bastien N, Lee SW, Krajden M, Brunham RC. Protective measures and human antibody response during an avian influenza H7N3 outbreak in poultry in British Columbia, Canada. CMAJ. 2007 Jan 2;176(1):47-53. doi: 10.1503/cmaj.060204. PMID 17200390
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_002421-I.html